CLINICAL TRIAL: NCT05411601
Title: Numerical Standard of Anthropomorphicity of Prosthetic Feet for Improvement of Amputee Performance
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: PolyOrth International (Industry)
Responsible Party: Sponsor
Other Study IDs: POI 012022
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Testing of Methodology of Attachment of External Foot Prothesis Based on Anthropomorphism Criteria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- C1: Subjects with socket-type attachment of their prostheses
  Interventions: Other: Methodology of attachment of external foot prothesis
- C2: Subjects with direct skeletal attachment
  Interventions: Other: Methodology of attachment of external foot prothesis

INTERVENTIONS:
Other: Methodology of attachment of external foot prothesis — establishing the methodology of specific measurements of attachment of external foot prothesis

SUMMARY:
The study concerns the testing of methodology of attachment of external foot prothesis based on anthropomorphism criteria

ELIGIBILITY:
Inclusion Criteria:

* Unilateral lower transtibial amputation
* Prosthetic user with socket type attachment (Cohort 1) or with direct skeletal attachment (Cohort 2) and be able to walk 50 meters independently,
* Between 18-60 years of age,
* Able to follow instructions,
* Able to provide consent.

Exclusion Criteria:

* problems on the residuum,
* Non-prosthetic user,
* Bilateral amputation,
* Self-reported pain levels greater than 4 out of 10 at study outset,
* Experienced a fall within the last 8 weeks before assessment,
* Mental illness or intellectual impairment compromising participant's ability to give informed consent,
* Injuries involving contralateral (intact) limb,
* Major uncorrected visual deficit,
* History of epilepsy or recurrent dizziness,

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Subjects 18-60 years old that underwent unilateral lower transtibial amputation
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Stiffness and the index of anthropomorphicity IAm | 30 days
  Range of ankle stiffnesses, including three prostheses currently recommended to patients with direct skeletal attachment
IAb of the selected prosthetic feet | 30 days
  To establish IAb of the selected prosthetic feet via biomechanical gait testing

IPD SHARING:
Plan to Share IPD: No